CLINICAL TRIAL: NCT02740478
Title: A Comparison of the Non-contact Reassure Device Measurement Accuracy of Respiration Rate With SOMNOScreen, When Measured on a Continuous Basis Whilst the Subjects Are Asleep
Brief Title: Reassure Device: Measurement Accuracy of Continuous Respiration Rate
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: D22105-107
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Accuracy of Respiration Rate Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteers: 20 volunteer subjects, no selection criteria

SUMMARY:
The aim of the trial is to prove that the Reassure10.5 GHz sensor is equivalent in performance to the SomnoScreen Plus RC in indicating the breathing rate of adult subjects over a number of hours when the subjects are lying still or in bed asleep

DETAILED DESCRIPTION:
Each recording comprised at least 2 hours duration. The subject was lying on a bed, wearing the SomnoScreen and with the Reassure on a bed-side table in the recommended position: at arm's length, pointing at the subject's upper torso.

The subject was asked to lie in set positions on the bed for 20 minutes at a time. The data was recorded continuously for the duration of the trial and so encompassed the acts of turning from one position to another and any minor movement made by the subject. If the subject fell asleep during the trial, they were only woken when it came time for the next position change.

Key Duration Remarks Supine >=20minutes Subject Lying on back Prone >=20minutes Subject Lying face down Facing Left >=20minutes Subject's Chest facing Reassure device Facing Right >=20minutes Subject's Back facing Reassure device Foetal Left >=20minutes Subject's Chest facing Reassure device Foetal Right >=20minutes Subject's Back facing Reassure device

ELIGIBILITY:
Inclusion Criteria:

* Willing Volunteer

Exclusion Criteria:

* Restless leg syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Quantity 20 volunteer subjects willing to undergo the trial: lying still for 2 hours, following a pre-scripted set on lying positions.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Phillips, MA, MSc, Principal Investigator — ResMed Sensor Technologies Ltd

IPD SHARING:
Plan to Share IPD: No
Device performance validation, only registered with Clinicaltrials.gov as it entailed human volunteers. No intent to publish

REFERENCES:
- [Background] Lim WS, Carty SM, Macfarlane JT, Anthony RE, Christian J, Dakin KS, Dennis PM. Respiratory rate measurement in adults--how reliable is it? Respir Med. 2002 Jan;96(1):31-3. doi: 10.1053/rmed.2001.1203. PMID 11863207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteer subjects recruited until quantity 20 had completed the study
Groups:
- Reassure 10.5 GHz Sensor Sleep Simulation: Volunteer subjects, willing to undergo the trial of lying still on a bed for 2 hours. The subject's position changed every 20 minutes so that a range of positions explored. Subjects' respiration rate measure by the non-contact Reassure device and compared to a SomnoScreen device that uses chest effort belts to record the respiration rate.
  Volunteers recruited until there were 20 that completed the study.
Period: Overall Study
Arm/Group | Reassure 10.5 GHz Sensor Sleep Simulation
Started | 21 (Volunteers recruited until quantity 20 completed the study)
Completed | 20 (One volunteer was very high BMI and uncomfortable lying still during the recordings: test stopped.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reassure 10.5 GHz Sensor Sleep Simulation
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  Ireland | 20

OUTCOME MEASURES:

1. Primary Outcome: Respiration Rate Comparability
Description: The respiration rate measured contemporaneously by the Reassure and the reference device, SomnoScreen, are compared on a second-by-second basis, over the whole recording duration. The difference between the two respiration rate measurements (the delta) for all 20 subjects' recordings are plotted on a normal distribution chart, giving 130,000 data points. The distribution chart reveals the mean difference between the two devices' measurements and the Standard Deviation (SD). The measure of success is if the 95% (ie 2SD) of the difference in the respiration rate indicated by the two devices (the delta) is less than 5 breaths per minute. This measure is derived from the peer review paper by Lim et al, cited in the References section
Time Frame: 2 hour recording
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Reassure 10.5 GHz Sensor Sleep Simulation
Number analyzed (Participants) | 20
breaths per minute | 0.4 (1.2)

ADVERSE EVENTS:
Time Frame: 2 hours during which the evaluation took place
Arm/Group | Reassure 10.5 GHz Sensor Sleep Simulation
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes